CLINICAL TRIAL: NCT06878222
Title: Iparomlimab and Tuvonralimab Combined With Paclitaxel and Cisplatin as Neoadjuvant Therapy for Cervical Cancer: a Phase 2 Umbrella Trial
Brief Title: Iparomlimab and Tuvonralimab Combined With Paclitaxel and Cisplatin as Neoadjuvant Therapy for CC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Keqin Hua, Director of Gynecological Oncology, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QIBA-CER-003
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancers
Keywords: cervical cancer; neoadjuvant therapy; Iparomlimab and Tuvonralimab; immunotherapy; fertility-preserving
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Neoadjuvant Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm1: locally advanced cervical cancer (Active Comparator): Patients with locally advanced cervical cancer classified as FIGO 2018 stages IB3, IIA2, IIB, or IIICr (lesion ≥4 cm, confirmed by MRI); histologically confirmed cervical squamous cell carcinoma, cervical adenocarcinoma, or cervical adenosquamous carcinoma；18-75 years old.
  Interventions: Drug: Neoadjuvant Chemotherapy; Drug: Immunotherapy; Procedure: Radical surgery
- Arm2: cervical cancer patients desiring fertility-preserving treatment (Active Comparator): Patients with cervical cancer classified as FIGO 2018 stages IB2, IB3 (lesion ≤6 cm), IIA1, or IIA2 (lesion ≤6 cm) who have a strong desire to preserve fertility； histologically confirmed cervical squamous cell carcinoma, cervical adenocarcinoma, or cervical adenosquamous carcinoma； 18-45 years old.
  Interventions: Drug: Neoadjuvant Chemotherapy; Drug: Immunotherapy; Procedure: Fertility-preserving surgery

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — paclitaxel, 135-175mg/m2, q3w, 3 cycles
Drug: Neoadjuvant Chemotherapy — cisplatin, 75-80mg/m2, q3w, 3 cycles
Drug: Immunotherapy — Iparomlimab and Tuvonralimab, 5mg/kg, q3w, 3cycles
Procedure: Radical surgery — After 3 cycles of neoadjuvant therapy, patients who achieved CR/PR will undergo radical hysterectomy plus lymphadenectomy
  Arms: Arm1: locally advanced cervical cancer
Procedure: Fertility-preserving surgery — After 3 cycles of neoadjuvant therapy, patients who achieved CR/PR will undergo Fertility-preserving surgery. For stage IB1/IB2 patients, conization or simple trachelectomy plus lymphadenectomy will be performed. For stage IIA1/IIA2 patients, radical trachelectomy plus lymphadenectomy will be performed.
  Arms: Arm2: cervical cancer patients desiring fertility-preserving treatment

SUMMARY:
Currently, the survival rate of locally advanced cervical cancer is low, posing a significant challenge in the treatment of cervical cancer. Radical chemoradiotherapy is considered the standard treatment for patients with locally advanced cervical cancer. However, 23.3% to 34.4% of patients still experience recurrence or subsequent metastasis. Radical surgery following neoadjuvant chemotherapy is an alternative to concurrent chemoradiotherapy, but it also has limitations: for approximately 9.8% to 30.6% of patients who do not respond to neoadjuvant chemotherapy, effective local treatment may be delayed. Additionally, more than 30% of patients still require adjuvant radiotherapy or chemoradiotherapy after surgery, significantly increasing the risk of complications. Therefore, there is an urgent need to explore alternative or improved treatment methods for neoadjuvant chemotherapy in locally advanced cervical cancer.

An increasing number of women are being diagnosed with cervical cancer during their childbearing years, many of whom have a desire to preserve their fertility. For selected patients with stage IB2 cervical cancer, options include abdominal radical trachelectomy or radical trachelectomy following neoadjuvant chemotherapy. However, compared to conservative surgeries such as conization or partial cervical resection, radical trachelectomy is associated with less favorable fertility rates and pregnancy outcomes, with significantly higher rates of infertility, miscarriage, and preterm birth. For patients with stage IB3 or IIA1-IIA2 cervical cancer, the current standard surgical approach is radical hysterectomy, which does not preserve fertility. Current research suggests that neoadjuvant chemotherapy can shrink tumor size, decrease lymph node and distant metastases, and reduce the need for postoperative adjuvant radiotherapy. This offers hope for young cervical cancer patients who wish to preserve fertility, as it may reduce tumor size, thereby allowing for less extensive fertility-sparing surgery, improving pregnancy outcomes, or even making fertility-sparing surgery a viable option.

In recent years, immunotherapy has gradually become a research hotspot in cancer treatment. Anti-PD-1/PD-L1 monoclonal antibodies, as a type of immunotherapy drug, have demonstrated promising anti-tumor efficacy and low side effects in clinical trials. Iparomlimab and Tuvonralimab is a novel therapeutic biological product targeting both PD-1 and CTLA-4. It is composed of two engineered monoclonal antibodies (anti-PD-1 and anti-CTLA-4) expressed in a fixed ratio and has shown significant efficacy in cervical cancer patients. Therefore, given the urgent need to improve neoadjuvant therapy for locally advanced cervical cancer and fertility-preserving neoadjuvant therapy for early-stage cervical cancer patients, this study is being conducted to explore and evaluate the efficacy and safety of Iparomlimab and Tuvonralimab combined with paclitaxel and cisplatin as neoadjuvant therapy for cervical cancer. Additionally, the study aims to investigate the relationship between tumor-related biomarkers and the risk of recurrence.

DETAILED DESCRIPTION:
In recent years, anti-PD-1/PD-L1 monoclonal antibodies, as a type of immunotherapy drug, have demonstrated promising anti-tumor efficacy in the treatment of cervical cancer patients. PD-1 (Programmed cell death protein 1) is a surface immune checkpoint protein that, by binding to its ligand PD-L1, inhibits the activation of T cells, thereby allowing tumor cells to evade immune system attacks. At the 2024 American Society of Clinical Oncology (ASCO) Annual Meeting, a phase II clinical study was reported on the use of immunotherapy (sintilimab) combined with paclitaxel and cisplatin as neoadjuvant therapy for locally advanced cervical cancer. The results showed that the primary endpoint, pathological complete response (pCR), was 32.6% (14/43), and the best response rate (residual tumor infiltration depth less than 3 mm) was 51.2% (22/43).

Iparomlimab and Tuvonralimab is a novel therapeutic biological product targeting both PD-1 and CTLA-4. It is composed of two engineered monoclonal antibodies (anti-PD-1 and anti-CTLA-4) expressed in a fixed ratio and produced as a single product from a single cell line. It offers the following advantages:

1. Dual immune targets of PD-1 and CTLA-4 monoclonal antibodies: The anti-PD-1 antibody relieves T cell killing inhibition, while the anti-CTLA-4 antibody relieves T cell activation inhibition, working synergistically to enhance efficacy.
2. Optimal 2:1 ratio of anti-PD-1 to anti-CTLA-4 antibodies: A dosing regimen of 5 mg/kg every 3 weeks ensures effective blood concentration, balancing efficacy and safety.
3. Flexible antibody subtype design: The anti-PD-1 antibody uses the IgG4 subtype, which lacks ADCC (antibody-dependent cellular cytotoxicity) effects and does not deplete effector T cells. The anti-CTLA-4 antibody uses the IgG1 subtype, which has ADCC effects and can eliminate regulatory T cells, further enhancing efficacy.
4. R255K mutation in the anti-CTLA-4 antibody: This mutation reduces the affinity of the anti-CTLA-4 antibody for the neonatal Fc receptor (FcRn), shortening its half-life to 1 week and lowering its blood concentration, thereby improving safety while maintaining efficacy.

Currently, Iparomlimab and Tuvonralimab for recurrent or metastatic cervical cancer as a second-line or later treatment has shown an objective response rate (ORR) of 33.8% and a progression-free survival (PFS) of 5.4 months, with a favorable safety profile. When combined with chemotherapy as first-line treatment for recurrent or metastatic cervical cancer, the ORR was 75.9%, PFS was 15.1 months, and immune-related adverse events occurred in 16.7% of cases. These results indicate that Iparomlimab and Tuvonralimab, both as monotherapy and in combination therapy, demonstrates significant anti-tumor activity and safety, suggesting that dual-target antibodies are effective for advanced cancer patients.

Therefore, given the urgent need to improve neoadjuvant therapy for locally advanced cervical cancer and neoadjuvant fertility-preserving therapy for early-stage cervical cancer, this study is being conducted to explore and evaluate the efficacy and safety of Iparomlimab and Tuvonralimab combined with paclitaxel and cisplatin as neoadjuvant therapy for locally advanced cervical cancer and fertility-preserving neoadjuvant therapy for cervical cancer. Additionally, the study aims to investigate the relationship between tumor-related biomarkers and the risk of recurrence, potentially offering new insights for optimizing fertility-preserving and non-preserving neoadjuvant therapies for cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed cervical squamous cell carcinoma, cervical adenocarcinoma, or cervical adenosquamous carcinoma.
2. -Arm 1 (Locally Advanced cervical cancer): Patients with locally advanced cervical cancer classified as FIGO 2018 stages IB3, IIA2, IIB, or IIICr (lesion ≥4 cm, confirmed by MRI).

   * Arm2 (cervical cancer patients desiring fertility-sparing treatment): Patients with cervical cancer classified as FIGO 2018 stages IB2, IB3 (lesion ≤6 cm), IIA1, or IIA2 (lesion ≤6 cm) who have a strong desire to preserve fertility.

     3）Planned to undergo surgical treatments of cervical cancer.

4) -Arm 1 (Locally Advanced cervical cancer): Age 18-75 years.

* Arm2 (cervical cancer patients desiring fertility-sparing treatment): Age 18-45 years.

  5) ECOG performance status score: 0-1. 6) No prior immunotherapy received by the participant. 7) Expected survival period ≥6 months. 8) Women of childbearing potential must agree to use contraception (e.g., intrauterine device, oral contraceptives, or condoms) during the study and for 6 months after the study ends. A negative serum or urine pregnancy test within 7 days before study enrollment is required, and the patient must not be breastfeeding.

  9) Adequate organ function as defined by the protocol, with test samples collected within 7 days before the start of study treatment.

  10) Participants voluntarily join the study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Histological subtypes or disease stages other than those permitted in inclusion criteria 1) and 2).
2. Severe hypersensitivity (≥ Grade 3) to cisplatin, paclitaxel, iparomlimab and tuvonralimab, and/or any of their excipients.
3. Participation in another clinical trial within 4 weeks prior to enrollment.
4. Administration of inactivated vaccines within 30 days before the first study treatment or planned vaccination during the study period.
5. Treatment with systemic immunostimulants, colony-stimulating factors, interferons, interleukins, or combination vaccines within 6 weeks or 5 half-lives (whichever is shorter) before the first dose.
6. Diagnosis of immunodeficiency or chronic systemic steroid therapy (exceeding 10 mg prednisone equivalent per day) or any other form of immunosuppressive therapy within 7 days before the first dose.
7. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressive drugs) within the past 2 years.
8. History of (non-infectious) pneumonitis requiring steroid treatment or current (non-infectious) pneumonitis.
9. Active infection requiring systemic treatment.
10. Known history of HIV infection.
11. Known history of hepatitis B (defined as HBsAg reactivity) or active hepatitis C virus infection (defined as detectable HCV RNA [qualitative]).
12. Known history of active tuberculosis (TB; Mycobacterium tuberculosis).
13. Prior allogeneic tissue/solid organ transplantation.
14. Central nervous system metastases, such as brain metastases.
15. Uncontrolled pleural or peritoneal effusion.
16. Impaired mobility due to pathological fractures caused by bone metastases.
17. Insufficient bone marrow function (without transfusion within 14 days): a) Absolute neutrophil count (ANC) <1.5×10⁹/L;b) Platelets <100×10⁹/L; c) Hemoglobin <9 g/dL.
18. Liver abnormalities: a) ALT, AST, or ALP >2.5× upper limit of normal (ULN) without liver metastasis or >5×ULN with liver metastasis; b) Total bilirubin >1.5×ULN (>3×ULN in patients with Gilbert's syndrome); c) Decompensated cirrhosis (Child-Pugh class B or C); d) HBsAg-positive with HBV DNA ≥2000 IU/mL (patients with HBsAg-positive and HBV DNA <2000 IU/mL must receive at least 2 weeks of anti-HBV therapy before the first dose); e) HCV antibody-positive with detectable HCV RNA.
19. Kidney abnormalities: a) Serum creatinine >1.5×ULN or estimated creatinine clearance <60 mL/min using the Cockcroft-Gault formula; b) Urinalysis showing protein ≥++ and confirmed 24-hour urine protein >1.0 g; c) Renal failure requiring hemodialysis or peritoneal dialysis; d) History of nephrotic syndrome.
20. Bleeding risk: a) Coagulation abnormalities: Activated partial hromboplastin time (APTT) or thrombin time (TT) >1.5×ULN, or international normalized ratio (INR) >1.5 (>2.5 for patients requiring anticoagulation therapy); b) History of bleeding (e.g., hemoptysis), coagulation disorders, or current use of warfarin, aspirin, low-molecular-weight heparin, or other antiplatelet agents (except for aspirin ≤100 mg/d for prophylaxis); c) Any signs or history of bleeding diathesis, regardless of severity; d) Active gastrointestinal bleeding, evidenced by hematemesis, hematochezia, or melena within the past 3 months, without resolution confirmed by endoscopy or colonoscopy; e) Any CTCAE ≥ Grade 3 bleeding or hemorrhagic event within 4 weeks before the first dose.
21. Cardiovascular and cerebrovascular abnormalities: a) Any of the following within 12 months before the first dose: ≥ Grade 2 myocardial ischemia, yocardial infarction, arrhythmias, ≥ Grade 3 cardiac insufficiency, uncontrolled angina, coronary/peripheral artery bypass graft surgery, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack; b) Deep vein thrombosis or pulmonary embolism within 6 months before the first dose; c) Left ventricular ejection fraction (LVEF) <50% assessed by Doppler ultrasound; d) Average QTc interval corrected by Fridericia's formula (QTcF) (based on at least 3 consecutive ECG readings): ≥470 ms for females; e) Uncontrolled hypertension (at least 2 measurements showing systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg).
22. Other factors judged by the investigator as potentially affecting study results or leading to premature termination, such as alcoholism, drug abuse, other severe diseases (including mental illness) requiring concurrent treatment, significant laboratory abnormalities, or family/social factors that may compromise patient safety.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 9 weeks
  ORR measures the proportion of patients whose cervical cancer shows a complete response (CR) or partial response (PR) to neoadjuvant therapy in this study. Complete Response (CR) means total disappearance of all detectable tumors and partial Response (PR) means significant reduction in tumor size larger than 30% according to RECIST guidelines.
Pathological Complete Response (pCR) | 3 months
  Pathological Complete Response (pCR) refers to the absence of detectable cancer cells in the tissue removed during surgery after neoadjuvant therapy which is examined under a microscope by a pathologist.
changes in tumor-related biomarkers | 3 months

SECONDARY OUTCOMES:
OS (Overall Survival) | 2 years
DFS (Disease Free Survival) | 2 years
adverse events | 2 years

OTHER OUTCOMES:
Pregnancy rate | 2 years
infant survival rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Keqin Hua, Doctor, Principal Investigator — Gynecology and obstetrics hospital of fudan university
Locations (1):
- The Obstetrics & Gynecology Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No